CLINICAL TRIAL: NCT02718326
Title: A Phase 3, Double-Masked, Randomized Study of the Efficacy and Safety of Intravitreal Aflibercept Injection in Patients With Moderately Severe to Severe Nonproliferative Diabetic Retinopathy
Brief Title: Study of the Efficacy and Safety of Intravitreal (IVT) Aflibercept for the Improvement of Moderately Severe to Severe Nonproliferative Diabetic Retinopathy (NPDR)
Acronym: PANORAMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VGFTe-OD-1411; 2016-002639-14 (EudraCT Number)
Record Dates: First submitted 2016-03-20; First posted 2016-03-24 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Nonproliferative Diabetic Retinopathy
MeSH Terms: interventions — aflibercept; Injections; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dosing regimen 1 (Experimental): Participants will receive IVT aflibercept dosing regimen 1
  Interventions: Drug: Intravitreal aflibercept injection [IAI]
- Dosing regimen 2 (Experimental): Participants will receive IVT aflibercept dosing regimen 2
  Interventions: Drug: Intravitreal aflibercept injection [IAI]
- Dosing regimen 3 (Sham Comparator): Participants will receive matching sham injections
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: Intravitreal aflibercept injection [IAI]
  Other Names: EYLEA® (aflibercept) Injection; BAY86-5321
  Arms: Dosing regimen 1; Dosing regimen 2
Drug: Sham
  Arms: Dosing regimen 3

SUMMARY:
The primary objective of the study is to assess the efficacy of intravitreal (IVT) aflibercept compared to sham treatment in the improvement of moderately severe to severe nonproliferative diabetic retinopathy (NPDR).

The secondary objectives of the study are:

* To characterize the safety of IVT aflibercept in patients with moderately severe to severe NPDR
* To determine if IVT aflibercept will prevent the worsening of diabetic retinopathy and reduce the incidence of DME
* To determine the anatomic effects of IVT aflibercept in patients with moderately severe to severe NPDR

ELIGIBILITY:
Key Inclusion Criteria:

1. Men or women ≥18 years of age with type 1 or 2 diabetes mellitus who have moderately severe to severe nonproliferative diabetic retinopathy (NPDR) [(diabetic retinopathy severity scale (DRSS) levels 47 or 53)], confirmed by the central reading center, in whom panretinal photocoagulation (PRP) can be safely deferred for at least 6 months per the investigator
2. Best corrected visual acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) letter score in the study eye of ≥69 letters (approximate Snellen equivalent of 20/40 or better)

Key Exclusion Criteria:

1. Presence of diabetic macular edema (DME) threatening the center of the macula in the study eye
2. Evidence of retinal neovascularization on clinical examination or Fluorescein Angiography (FA)
3. Any prior focal or grid laser photocoagulation or any prior PRP in the study eye
4. Any prior systemic anti-vascular endothelial growth factor (VEGF) treatment or intravitreal (IVT) anti-VEGF treatment in the study eye
5. Any prior intraocular steroid injection in the study eye
6. Current anterior segment neovascularization (ASNV), vitreous hemorrhage, or tractional retinal detachment visible at the screening assessments in the study eye

Note: Other inclusion/ exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (85):
- United States (68):
  - Regeneron Study Site, Phoenix, Arizona
  - Regeneron Study Site, Tucson, Arizona
  - Regeneron Study Site, Arcadia, California
  - Regeneron Study Site, Beverly Hills, California
  - Regeneron Study Site, Encino, California
  - Regeneron Study Site, Fullerton, California
  - Regeneron Study Site, La Jolla, California
  - Regeneron Study Site, Mountain View, California
  - Regeneron Study Site, Oakland, California
  - Regeneron Study Site, Oceanside, California
  - Regeneron Study Site, Sacramento, California
  - Regeneron Study Site, Colorado Springs, Colorado
  - Regeneron Study Site, Golden, Colorado
  - Regeneron Study Site, New London, Connecticut
  - Regeneron Study Site, Altamonte Springs, Florida
  - Regeneron Study Site, Deerfield Beach, Florida
  - Regeneron Study Site, Fort Myers, Florida
  - Regeneron Study Site, Lakeland, Florida
  - Regeneron Study Site, Largo, Florida
  - Regeneron Study Site, Melbourne, Florida
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, Orlando, Florida
  - Regeneron Study Site, Plantation, Florida
  - Regeneron Study Site, Tallahassee, Florida
  - Regeneron Study Site, Tampa, Florida
  - Regeneron Study Site, Winter Haven, Florida
  - Regeneron Study Ssites, Marietta, Georgia
  - Regeneron study Site, Tucker, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site, Oak Forest, Illinois
  - Regeneron Study Site, Indianapolis, Indiana
  - Regeneron Study Site, New Albany, Indiana
  - Regeneron Study Site, Lexington, Kentucky
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Siste, Baltimore, Maryland
  - Regeneron Study Site, Hagerstown, Maryland
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Henderson, Nevada
  - Regeneron Study Site, Bloomfield, New Jersey
  - Regeneron Study Site, Albuquerque, New Mexico
  - Regeneron Study Site, Asheville, North Carolina
  - Regeneron Study Site, Charlotte, North Carolina
  - Regeneron Study Site, Columbus, Ohio
  - Regeneron Study Site, Oklahoma City, Oklahoma
  - Regeneron Study Site, Medford, Oregon
  - Regeneron Study Site, Kingston, Pennsylvania
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Florence, South Carolina
  - Regeneron Study Site, Ladson, South Carolina
  - Regeneron Study Site, West Columbia, South Carolina
  - Regeneron Study Site, Rapid City, South Dakota
  - Regeneron Study Site, Chattanooga, Tennessee
  - Regeneron Study Site, Germantown, Tennessee
  - Regeneron Study Site, Nashville, Tennessee
  - Regeneron Study Site, Abilene, Texas
  - Regeneron Study Site 1, Austin, Texas
  - Regeneron Study Site 2, Austin, Texas
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Harlingen, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, San Antonio, Texas
  - Regeneron Study Site, The Woodlands, Texas
  - Regeneron Study Site, Willow Park, Texas
  - Regeneron Study Site, Salt Lake City, Utah
  - Regeneron Study Site, Burlington, Vermont
  - Regeneron Study Site, Fairfax, Virginia
  - Regeneron Study Site, Spokane, Washington
  - Regeneron Study Site, Morgantown, West Virginia
- Germany (3):
  - Regeneron Study Site, Marburg, Hesse
  - Regeneron Study Site, Münster, North Rhine-Westphalia
  - Regeneron Study Site, Leipzig, Saxony
- Hungary (4):
  - Regeneron Study Site, Szeged, Csongrád megye
  - Regeneron Study Site, Debrecen, Hajdú-Bihar
  - Regeneron Study Site, Budapest, Pest County
  - Regeneron Study Site, Zalaegerszeg, Zala County
- Japan (6):
  - Regeneron Study Site, Asahikawa, Hokkaido
  - Regeneron Study Site, Amagasaki, Hyōgo
  - Regeneron Study Site, Matsumoto, Nagano
  - Regeneron Study Site, Chiyoda City, Tokyo
  - Regeneron Study Site, Kagoshima
  - Regeneron Study Site, Nagasaki
- Puerto Rico (2):
  - Regeneron Study Site, Arecibo
  - Regeneron Study Site, San Juan
- United Kingdom (2):
  - Regeneron Study Site, Camberley, Surrey
  - Regeneron Study Site, London

REFERENCES:
- [Derived] Brown DM, Wykoff CC, Boyer D, Heier JS, Clark WL, Emanuelli A, Higgins PM, Singer M, Weinreich DM, Yancopoulos GD, Berliner AJ, Chu K, Reed K, Cheng Y, Vitti R. Evaluation of Intravitreal Aflibercept for the Treatment of Severe Nonproliferative Diabetic Retinopathy: Results From the PANORAMA Randomized Clinical Trial. JAMA Ophthalmol. 2021 Sep 1;139(9):946-955. doi: 10.1001/jamaophthalmol.2021.2809. PMID 34351414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study was conducted in the following countries between 29 Mar 2016 and 07 Aug 2017: Germany, Hungary, Japan, the United Kingdom, and the United States. A total of 759 participants were screened.
Pre-assignment Details: Out of 759, 402 participants were randomized to receive 1 of 3 treatment groups in a 1:1:1 ratio stratified based on their Diabetic Retinopathy Severity Scale (DRSS) score (level 47 vs. level 53). Only 1 eye was selected as the study eye.
Units Other Than Participants: Eyes
Groups:
- Sham Treatment: All participants received sham injections in the study eye every 4 weeks (Q4) to week 16 (after 5 initial monthly sham injections), followed by sham injections Q8 to week 96.
- Intravitreal Aflibercept Injection (IAI) 2Q16: All participants received a 2 milligram (mg) Intravitreal Aflibercept Injection (IAI) in the study eye every 16 weeks (2Q16) (after 3 initial monthly doses and one 8-week interval) to week 96.
- Intravitreal Aflibercept Injection (IAI) 2Q8: All participants received 2 mg IAI in the study eye every 8 weeks (2Q8) from day 1 up to week 48 (after 5 initial monthly doses), followed by a flexible treatment regimen with IAI 2 mg to week 96.
Period: Overall Study
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8
Started | 133; 133 Eyes | 135; 135 Eyes | 134; 134 Eyes
Completed Week 52 | 109; 109 Eyes | 122; 122 Eyes | 124; 124 Eyes
Completed (Week 100 (End of Study)) | 97; 97 Eyes | 111; 111 Eyes | 112; 112 Eyes
Not Completed | 36; 36 Eyes | 24; 24 Eyes | 22; 22 Eyes
Not completed — Adverse Event | 4 | 9 | 0
Not completed — Death | 8 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 9 | 6
Not completed — Lost to Follow-up | 18 | 5 | 14
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received any study treatment as assigned at baseline (as randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8 | Total
Number analyzed (Participants) | 133 | 135 | 134 | 402
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.8 (10.31) | 55.4 (11.13) | 55.8 (10.19) | 55.7 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 60 | 53 | 177
  Male | 69 | 75 | 81 | 225
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 97 | 93 | 264
  Not Hispanic or Latino | 58 | 37 | 41 | 136
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 4 | 6
  Asian | 4 | 12 | 7 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 13 | 16 | 12 | 41
  White | 107 | 99 | 104 | 310
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 8 | 5 | 5 | 18
Baseline Diabetic Retinopathy Severity Score (DRSS) [Count of Participants; unit: Participants] — The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached).
  Participants
    Level 47 (Moderately Severe) | 99 | 102 | 101 | 302
    Level 53 (Severe) | 34 | 33 | 33 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Improved by ≥2 Steps From Baseline in the Diabetic Retinopathy Disease Severity Scale (DRSS) Score at Week 24 in the Combined 2Q16 and 2Q8 Groups
Description: The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached). Here, DRSS describes severity level 47 (moderately severe NPDR) and level 53 (severe NPDR) at week 24 from baseline.
Time Frame: At Week 24
Population: FAS included all randomized participants who received any study treatment as assigned at baseline (as randomized). The missing data were imputed using last observation carried forward (LOCF) method.
Measure: Number; unit: Percentage of participants
Groups:
- IAI 2 mg Groups Combined (2Q16 & 2Q8): IAI 2Q16: Participants received a 2 milligram (mg) Intravitreal Aflibercept Injection (IAI) in the study eye every 16 weeks (2Q16) (after 3 initial monthly doses and one 8-week interval) to week 96; IAI 2Q8: Participants received 2 mg IAI in the study eye every 8 weeks (2Q8) from day 1 up to week 48 (after 5 initial monthly doses), followed by a flexible treatment regimen with IAI 2 mg to week 96.
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8 | IAI 2 mg Groups Combined (2Q16 & 2Q8)
Number analyzed (Participants) | 133 | 135 | 134 | 269
Percentage of participants | 6.0 | 61.5 | 55.2 | 58.4
Statistical Analysis 1: Comparison: Sham Treatment vs IAI 2 mg Groups Combined (2Q16 & 2Q8); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; percentage difference = 52.3, 95% CI 2-sided [45.2 to 59.5]

2. Primary Outcome: Percentage of Participants With a ≥ 2-step Change at Week 52 in Diabetic Retinopathy Severity Scale (DRSS) From Baseline
Description: The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached). Here, DRSS describes severity level 47 (moderately severe NPDR) and level 53 (severe NPDR) at week 52 from baseline.
Time Frame: At Week 52
Population: FAS included all randomized participants who received any study treatment as assigned at baseline (as randomized). The missing data were imputed using LOCF method.
Measure: Number; unit: Percentage of participants
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8
Number analyzed (Participants) | 133 | 135 | 134
Percentage of participants | 15.0 | 65.2 | 79.9
Statistical Analysis 1: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; percentage difference = 50.1, 95% CI 2-sided [40.1 to 60.1]
Statistical Analysis 2: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q8; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; percentage difference = 64.8, 95% CI 2-sided [55.8 to 73.9]

3. Secondary Outcome: Percentage of Participants Who Developed a Vision-Threatening Complication Due to Diabetic Retinopathy at Week 52
Description: Vision-threatening complications are defined as the composite outcome of proliferative diabetic retinopathy (PDR) (inclusive of participants who have vitreous hemorrhage or tractional retinal detachment believed to be due to PDR) and anterior segment neovascularization (ASNV) (participants with neovascularization of the iris [at least 2 cumulative clock hours], and/or definitive neovascularization of the iridocorneal angle).
Time Frame: At Week 52
Population: FAS included all randomized participants who received any study treatment as assigned at baseline (as randomized).
Measure: Number; unit: Percentage of participants
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8
Number analyzed (Participants) | 133 | 135 | 134
Percentage of participants | 20.3 | 3.7 | 3.0
Statistical Analysis 1: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q8; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; percentage difference = -17.3, 95% CI 2-sided [-24.7 to -9.9]
Statistical Analysis 2: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; percentage difference = -16.6, 95% CI 2-sided [-24.2 to -9.1]

4. Secondary Outcome: Percentage of Participants Who Developed Central Involved-Diabetic Macular Edema (CI-DME) at Week 52
Description: The percentage of participants who developed CI-DME at week 52 were reported.
Time Frame: At Week 52
Population: FAS included all randomized participants who received any study treatment as assigned at baseline (as randomized).
Measure: Number; unit: Percentage of participants
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8
Number analyzed (Participants) | 133 | 135 | 134
Percentage of participants | 25.6 | 6.7 | 8.2
Statistical Analysis 1: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q8; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; percentage difference = -17.3, 95% CI 2-sided [-26.2 to -8.5]
Statistical Analysis 2: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; percentage difference = -18.9, 95% CI 2-sided [-27.5 to -10.4]

5. Secondary Outcome: Time to Development of Any Neovascular Vision Threatening Complication (PDR/ASNV) Through Week 52
Description: Vision-threatening complication (VTC) is defined as the composite outcome of proliferative diabetic retinopathy (PDR) (inclusive of participants who have vitreous hemorrhage or tractional retinal detachment believed to be due to PDR) and anterior segment neovascularization (ASNV) (participants with neovascularization of the iris [at least 2 cumulative clock hours], and/or definitive neovascularization of the iridocorneal angle). Vision Threatening Complications include PDR/ASNV identified by investigators and Diabetic Retinopathy Scale Score (DRSS) >61.
Time Frame: Baseline through week 52 (day 365)
Population: FAS included all randomized participants who received any study treatment as assigned at baseline (as randomized). Participants who did not have an event were censored at their last visit at or before the week 52 visit.
  Here, the value "NA" = Not evaluable due to small number of VTC events.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8
Number analyzed (Participants) | 133 | 135 | 134
Days | NA [371 to NA] — NA = Not evaluable due to small number of VTC events | NA [NA to NA] — NA = Not evaluable due to small number of VTC events | NA [NA to NA] — NA = Not evaluable due to small number of VTC events

6. Secondary Outcome: Time to Development of Central Involved-Diabetic Macular Edema (CI-DME) Through Week 52
Description: Time to develop Central Involved-Diabetic Macular Edema (CI-DME) through week 52 reported.
Time Frame: Baseline through week 52 (day 365)
Population: FAS included all randomized participants who received any study treatment as assigned at baseline (as randomized). Participants who did not have an event were censored at their last visit, at or before the week 52 visit. Here, the value "NA" = Not evaluable due to small number of CI-DME events.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8
Number analyzed (Participants) | 133 | 135 | 134
Days | NA [333 to NA] — NA = Not evaluable due to small number of CI-DME events | NA [NA to NA] — NA = Not evaluable due to small number of CI-DME events | NA [NA to NA] — NA = Not evaluable due to small number of CI-DME events

7. Secondary Outcome: Percentage of Participants Who Received Panretinal Photocoagulation (PRP), Inclusive of Participants Undergoing Vitrectomy With Endolaser, at Week 52
Description: The percentage of participants who received panretinal photocoagulation (PRP), inclusive of participants undergoing vitrectomy with endolaser, at week 52 were reported.
Time Frame: At Week 52
Population: FAS included all randomized participants who received any study treatment as assigned at baseline (as randomized).
Measure: Number; unit: Percentage of participants
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8
Number analyzed (Participants) | 133 | 135 | 134
Percentage of participants | 6.8 | 0.7 | 0.7
Statistical Analysis 1: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q8; Test type: Superiority; p = 0.0096, Cochran-Mantel-Haenszel; percentage difference = -6.0, 95% CI 2-sided [-10.5 to -1.5]
Statistical Analysis 2: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q16; Test type: Superiority; p = 0.0089, Cochran-Mantel-Haenszel; percentage difference = -6.0, 95% CI 2-sided [-10.5 to -1.6]

8. Secondary Outcome: Area Under the Curve (AUC) for Change From Baseline in Best Corrected Visual Acuity (BCVA) at Week 52
Description: The area under the curve (AUC) is the area under the best corrected visual acuity (BCVA) versus time curve from baseline to week 52. Visual function of the study eye was assessed at a distance of 4 meters at every study visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. BCVA scale range is 0 (worst) to 100 (best).
Time Frame: At week 52
Population: AUC was calculated as a weighted average based on total AUC (using the trapezoidal rule) divided by total duration in days. FAS included all randomized participants who received any study treatment as assigned at baseline (as randomized).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8
Number analyzed (Participants) | 133 | 135 | 134
scores on a scale | 0.5 (3.01) | 1.7 (3.50) | 1.3 (3.49)
Statistical Analysis 1: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q8; Test type: Superiority; p = 0.0529, ANOVA; Estimate for contrast = 0.80, 95% CI 2-sided [-0.01 to 1.60]
Statistical Analysis 2: Comparison: Sham Treatment vs Intravitreal Aflibercept Injection (IAI) 2Q16; Test type: Superiority; p = 0.0057, ANOVA; Estimate for contrast = 1.14, 95% CI 2-sided [0.33 to 1.94]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to week 100 regardless of seriousness or relationship to investigational product
Description: Reported adverse events are treatment-emergent adverse events (TEAEs) which are AEs that developed/worsened from baseline (day1) up to end of study (week 100).
Arm/Group | Sham Treatment | Intravitreal Aflibercept Injection (IAI) 2Q16 | Intravitreal Aflibercept Injection (IAI) 2Q8 | IAI 2 mg Groups Combined (2Q16 & 2Q8)
All-Cause Mortality (participants affected / at risk) | 8/133 | 1/135 | 3/134 | 4/269
Serious Adverse Events (participants affected / at risk) | 38/133 | 38/135 | 47/134 | 85/269
Other Adverse Events (participants affected / at risk) | 104/133 | 104/135 | 106/134 | 210/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Treatment (N=133) | Intravitreal Aflibercept Injection (IAI) 2Q16 (N=135) | Intravitreal Aflibercept Injection (IAI) 2Q8 (N=134) | IAI 2 mg Groups Combined (2Q16 & 2Q8) (N=269)
Coronary artery disease (Cardiac disorders) | 1 (1) | 5 (5) | 4 (4) | 9 (9)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 5 (6) | 7 (8)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 3 (5) | 6 (8)
Diabetic foot infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocephalus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (5) | 1 (5)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced Fellow Eye (Eye disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Diabetic retinal oedema Fellow Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Macular fibrosis Fellow Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Macular hole Fellow Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retinal vein occlusion Fellow Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Visual impairment Fellow Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous adhesions Fellow Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous haemorrhage Fellow Eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cataract Fellow Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iris neovascularisation Fellow Eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cystoid macular oedema Study Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Visual acuity reduced Study Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous haemorrhage Study Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetic retinopathy Study Eye (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Iris neovascularisation Study Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal neovascularisation Study Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture Study Eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Treatment (N=133) | Intravitreal Aflibercept Injection (IAI) 2Q16 (N=135) | Intravitreal Aflibercept Injection (IAI) 2Q8 (N=134) | IAI 2 mg Groups Combined (2Q16 & 2Q8) (N=269)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5) | 7 (7) | 12 (12)
Nausea (Gastrointestinal disorders) | 8 (9) | 5 (5) | 6 (14) | 11 (19)
Bronchitis (Infections and infestations) | 7 (7) | 9 (10) | 5 (5) | 14 (15)
Cellulitis (Infections and infestations) | 6 (6) | 5 (10) | 7 (7) | 12 (17)
Influenza (Infections and infestations) | 8 (8) | 10 (12) | 4 (4) | 14 (16)
Nasopharyngitis (Infections and infestations) | 15 (16) | 11 (16) | 11 (12) | 22 (28)
Urinary tract infection (Infections and infestations) | 16 (22) | 12 (13) | 11 (13) | 23 (26)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 5 (7) | 8 (11) | 13 (18)
Blood glucose increased (Investigations) | 7 (8) | 3 (3) | 7 (7) | 10 (10)
Glycosylated haemoglobin increased (Investigations) | 7 (7) | 9 (9) | 9 (9) | 18 (18)
Diabetes mellitus (Metabolism and nutrition disorders) | 13 (15) | 11 (11) | 8 (8) | 19 (19)
Headache (Nervous system disorders) | 2 (2) | 7 (9) | 8 (8) | 15 (17)
Hypertension (Vascular disorders) | 25 (28) | 28 (32) | 20 (23) | 48 (55)
Blepharitis Fellow Eye (Eye disorders) | 1 (1) | 3 (3) | 7 (7) | 10 (10)
Cataract Fellow Eye (Eye disorders) | 4 (4) | 9 (9) | 4 (4) | 13 (13)
Conjunctival haemorrhage Fellow Eye (Eye disorders) | 6 (7) | 5 (14) | 8 (14) | 13 (28)
Diabetic retinal oedema Fellow Eye (Eye disorders) | 19 (25) | 17 (24) | 23 (27) | 40 (51)
Diabetic retinopathy Fellow Eye (Eye disorders) | 12 (13) | 13 (14) | 10 (10) | 23 (24)
Macular oedema Fellow Eye (Eye disorders) | 4 (4) | 7 (7) | 6 (6) | 13 (13)
Retinal exudates Fellow Eye (Eye disorders) | 8 (9) | 2 (2) | 6 (7) | 8 (9)
Vitreous haemorrhage Fellow Eye (Eye disorders) | 4 (4) | 8 (12) | 3 (3) | 11 (15)
Blepharitis Study Eye (Eye disorders) | 1 (1) | 2 (2) | 7 (7) | 9 (9)
Cataract Study Eye (Eye disorders) | 5 (5) | 8 (8) | 8 (8) | 16 (16)
Conjunctival haemorrhage Study Eye (Eye disorders) | 8 (14) | 18 (27) | 25 (34) | 43 (61)
Diabetic retinal oedema Study Eye (Eye disorders) | 43 (54) | 14 (22) | 19 (25) | 33 (47)
Diabetic retinopathy Study Eye (Eye disorders) | 22 (25) | 3 (4) | 5 (5) | 8 (9)
Eye pain Study Eye (Eye disorders) | 6 (8) | 11 (13) | 5 (5) | 16 (18)
Retinal exudates Study Eye (Eye disorders) | 6 (7) | 5 (5) | 9 (9) | 14 (14)
Vitreous detachment Study Eye (Eye disorders) | 4 (4) | 7 (7) | 7 (9) | 14 (16)
Vitreous floaters Study Eye (Eye disorders) | 3 (3) | 7 (8) | 13 (13) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT02718326/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT02718326/SAP_001.pdf